CLINICAL TRIAL: NCT05697900
Title: Creatine Monohydrate Versus Creatine Hydrochloride on Strength and Body Composition in Elite Team-Sport Athletes: A Three-arm Placebo-controlled Randomized Clinical Trial
Brief Title: Creatine Monohydrate Versus Creatine Hydrochloride on Strength and Body Composition in Elite Team-Sport Athletes
Acronym: CrM_CrHCl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dynamical Business and Science Society - DBSS International SAS (Network)
Collaborators: INDEPORTES Antioquia (Unknown); CES University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Acta161_N°994
Record Dates: First submitted 2022-12-31; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Healthy Lifestyle
Keywords: Creatine; Strength; Body Composition; Athletic performance; Nutritional supplementation
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Intervention Model Description: This was a double-blinded placebo-controlled repeated-measures randomized clinical trial in elite team-sport athletes with three arms in parallel.
Who Masked: Participant, Investigator
Masking Description: This was a double-blinded clinical trial since participants and those assessing the outcomes were blinded to the intervention. All groups were given small metallic plastic bags with five grams of powder identical in size, shape, and color but the placebo contained maltodextrin (Tecnas S.A., Medellín, Colombia).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Creatine monohydrate (Active Comparator): 5 g of creatine monohydrate per day for eight weeks
  Interventions: Dietary Supplement: Creatine Monohydrate
- Creatine hydrochloride (Experimental): 5 g of creatine hydrochloride per day for eight weeks
  Interventions: Dietary Supplement: Creatine Hydrochloride
- Placebo (Placebo Comparator): 5 g of maltodextrin per day for eight weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine Monohydrate — The CrM group supplemented the diet with five grams of micronized creatine monohydrate per day for eight weeks. The CrM supplement was fully dissolved in ≈500 mL of water and drank immediately after each training session (in the morning on non-training days).
  Arms: Creatine monohydrate
Dietary Supplement: Placebo — A placebo group intakes five grams of maltodextrin daily throughout the study. The placebo supplement was fully dissolved in ≈500 mL of water and drank immediately after each training session (in the morning on non-training days).
  Arms: Placebo
Dietary Supplement: Creatine Hydrochloride — The Cr-HCl group supplemented the diet with five grams of micronized creatine monohydrate per day for eight weeks. The Cr-HCl supplement was fully dissolved in ≈500 mL of water and drank immediately after each training session (in the morning on non-training days).
  Arms: Creatine hydrochloride

SUMMARY:
A triple-arm double-blinded placebo-controlled repeated-measures randomized clinical trial in Colombian elite team-sport athletes. The aim is to evaluate the effects on strength-related parameters and body composition after eight weeks of supplementation with creatine monohydrate (CrM) and creatine hydrochloride (Cr-HCl). The study will be reported following the Consolidated Standards of Reporting Trials (CONSORT) extension to Multi-Arm Parallel-Group Randomized Trials. All variables will be measured at baseline and after eight weeks.

DETAILED DESCRIPTION:
Creatine monohydrate (CrM) is the most studied nutritional supplement and, therefore, one of the most popular ergogenic nutritional aids for athletes. Studies have shown that CrM supplementation increases intramuscular creatine concentrations which enhances exercise performance and improves body composition in different populations (from young athletes to older adults).

It is important to note that the U.S. Food and Drug Administration (FDA) have recognized CrM as a safe ingredient (Generally Recognized as Safe, GRAS - No. GRN 000931). In spite of this, other forms such as creatine chloride (Cr-HCl) have been marketed as a more bioavailable sources of creatine. Since there are not studies that rigorously compare the effects of CrM versus Cr-HCl on physical performance and body composition, the aim of this study is to evaluate the effects of a 8-week supplementation protocol with the two forms of creatine (comparing to placebo) on neuromuscular strength and body composition in Colombian elite team-sport athletes.

ELIGIBILITY:
Inclusion Criteria:

* Practicing team sports at the competitive level (handball and softball)
* Having at least one year of competitive sports training experience (including strength training at least three times a week),
* Being attended at INDEPORTES Antioquia.

Exclusion Criteria:

* Those who do not wish to participate voluntarily (do not sign informed consent),
* Those who were taking nutritional supplements (including creatine) eight weeks prior to the start of the study,
* Those who had a diagnosed pathology or health issues.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Lower-limb muscle power | Eight weeks
  Countermovement and drop jump will be performed on contact mat (height in centimeters and time of flight in seconds)
Neuromuscular strength | Eight weeks
  The load-velocity profile in squat and bench press exercises will be obtained with a linear position transducer (load in kilograms versus mean propulsive velocity in meters per second).
Upper-limb muscle strength | Eight weeks
  Maximal shoulder external and internal strength will be measure with a isokinetic dynamometer.

SECONDARY OUTCOMES:
Body composition | Eight weeks
  Body composition was measured using dual-energy x-ray absorptiometry. Fat mass and lean mass in kilograms were reported.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Rojas-Jaramillo, PhD, Study Director — INDEPORTES Antioquia; Diego A Bonilla, PhD, Study Chair — DBSS International SAS
Locations (1):
- INDEPORTES Antioquia, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kreider RB, Jager R, Purpura M. Bioavailability, Efficacy, Safety, and Regulatory Status of Creatine and Related Compounds: A Critical Review. Nutrients. 2022 Feb 28;14(5):1035. doi: 10.3390/nu14051035. PMID 35268011
- [Background] Bonilla DA, Kreider RB, Stout JR, Forero DA, Kerksick CM, Roberts MD, Rawson ES. Metabolic Basis of Creatine in Health and Disease: A Bioinformatics-Assisted Review. Nutrients. 2021 Apr 9;13(4):1238. doi: 10.3390/nu13041238. PMID 33918657
- [Background] Juszczak E, Altman DG, Hopewell S, Schulz K. Reporting of Multi-Arm Parallel-Group Randomized Trials: Extension of the CONSORT 2010 Statement. JAMA. 2019 Apr 23;321(16):1610-1620. doi: 10.1001/jama.2019.3087. PMID 31012939